CLINICAL TRIAL: NCT03727503
Title: Ability of a New PPV Smartphone Application to Predict Fluid Responsiveness in Cardiac Surgical Patients in the ICU
Brief Title: Casptesia Versus PICCO in Cardiac Surgical Patients in the ICU
Acronym: Capstesia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Logisitic problem
Sponsor: Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Alexandre Joosten, MD PhD, Principal Investigator, Erasme University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P2018/487
Record Dates: First submitted 2018-10-29; First posted 2018-11-01 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Surgery

STUDY DESIGN:
Intervention Model Description: Agreement and precision between two methods to measure pulse pressure variation (PPV)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- group/cohort (Other): operated patients from cardiac surgery. Once they arrived in the ICU, we will measure PPV with the capstesia and the PICCO device at baseline, and after a volume expansion of 500 ml of crystalloid.
  Interventions: Other: PPV from the capstesia

INTERVENTIONS:
Other: PPV from the capstesia — we will challenge the application by doing 2 maneuvers: the first one is to increase the PEEP level from 5 to 15 cmH2O and the second one is the infusion of a mini-fluid challenge (100 ml) followed by the other 400 ml.

SUMMARY:
The goal of this study is to assess the ability of a new smartphone PPV app to predict fluid responsiveness in cardiac surgical patients in the Intensive care unit (in the postoperative period)

DETAILED DESCRIPTION:
Pulse pressure variation (PPV) remains a good predictor of fluid responsiveness in the ICU in ventilated and sedated patients. However, PPV can be time-consuming to calculate (manual determination), is not always displayed on monitoring screens nor reliable through visual assessment and needs additional often costly devices to be displayed. A new Android application (Captesia) automatically calculates the PPV utilizing a digital photograph of the arterial waveform from the monitor. The application determines the PPV by selecting peaks and troughs of the arterial curve.

ELIGIBILITY:
Inclusion Criteria:

* adults patients ( >18 years)
* Patients scheduled for cardiac surgery
* equipped with a femoral arterial catheter and the PICCO device

Exclusion Criteria:

* Atrial fibrillation
* severe cardiac dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
PPV measure | baseline
  PPV before with after 2 maneuvers which modify PPV (increase PEEP level and mini-fluid challenge)
PPV measure | 1 minute after the end of volume expansion
  PPV before with after 2 maneuvers which modify PPV (increase PEEP level and mini-fluid challenge)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Joosten, M.D, Principal Investigator — ERASME
Locations (1):
- Erasme Hospital, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided